CLINICAL TRIAL: NCT05291806
Title: Second Meal Effects of a Wholegrain Cereal Product on Blood Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TSP2201
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-03

CONDITIONS: Blood Glucose Response

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference (Placebo Comparator)
  Interventions: Other: Reference Product
- Whole cereal kernels Dose A (Active Comparator)
  Interventions: Other: Wholegrain product Dose A
- Whole cereal kernels Dose B (Active Comparator)
  Interventions: Other: Wholegrain product Dose B
- Cut cereal kernels Dose A (Active Comparator)
  Interventions: Other: Wholegrain product Dose A, cut kernels

INTERVENTIONS:
Other: Reference Product — This intervention is based on white rice.
  Arms: Reference
Other: Wholegrain product Dose A — This wholegrain intervention contains whole cereal kernels.
  Arms: Whole cereal kernels Dose A
Other: Wholegrain product Dose B — This wholegrain intervention contains whole cereal kernels.
  Arms: Whole cereal kernels Dose B
Other: Wholegrain product Dose A, cut kernels — This wholegrain intervention contains cut cereal kernels.
  Arms: Cut cereal kernels Dose A

SUMMARY:
The aim of this study is to investigate second meal effects of a wholegrain cereal product on blood glucose response. The wholegrain cereal product will be consumed in the evening and blood glucose analyzed after a standardized breakfast meal the following morning.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 35 to 65 years of age
2. BMI 18.5-29.9 kg/m2
3. Agree to maintain consistent dietary habits and physical activity levels for the duration of the study.
4. Healthy as determined by medical history and information provided by the volunteer.
5. Willingness to complete questionnaires and follow instructions associated with the study and to complete all visits.
6. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Elevated fasting blood glucose (above 6.1 mmol/L at fasting on visit 1, 2, 3 or 4)
2. Women who are pregnant or breast feeding
3. Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the QI
4. Use of medication, over-the-counter medication, natural health products or dietary supplements/probiotics that may affect glucose metabolism is prohibited during this study. Significance to be assessed by the QI. Participants who are taking allowed prescribed medications must agree to maintain their current method and dosing regimen during the course of the study unless other is recommended by their physician.
5. Known Type I or Type II diabetes, including women who previously have had gestational diabetes.
6. Use of antibiotics within 2 weeks of enrollment
7. Metabolic diseases and/or chronic gastrointestinal diseases (IBS, Crohns etc.)
8. Allergy to ingredients included in investigational product, reference, or standardized meal
9. Participants restricted to a vegetarian or vegan diet
10. Intolerance to gluten
11. Individuals who are averse to venous catheterization or capillary blood sampling
12. Currently active smokers (or using other tobacco products, and e-cigarettes)
13. Unstable medical conditions as determined by QI
14. Participation in other clinical research trials
15. Individuals who are cognitively impaired and/or who are unable to give informed consent
16. Acute infection
17. Any other condition which in the QI's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual

    -

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Postprandial capillary blood glucose iAUC (0-120 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in capillary blood glucose between wholegrain products and reference in the total incremental area under the curve iAUC(0-120 min) after the standardized breakfast meal.

SECONDARY OUTCOMES:
Postprandial capillary blood glucose Cmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in capillary blood glucose between wholegrain products and reference in 2-hour Cmax(0-120 min) (maximum concentration) after the breakfast meal.
Postprandial capillary blood glucose Tmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in capillary blood glucose between wholegrain products and reference in 2-hour Tmax(0-120 min) (the time to maximum concentration) after the breakfast meal.
Fasting capillary blood glucose | Outcome measures will be assessed just before the standardized meal is consumed.
  The change in fasting capillary blood glucose the morning after consuming either wholegrain products or reference.
Postprandial capillary blood glucose iAUC (0-60 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in capillary blood glucose between wholegrain products and reference in the 1-hour incremental area under the curve iAUC(0-60 min) after the standardized breakfast meal.
Postprandial capillary blood glucose 2-hour iPeak(0-120 min) (incremental maximum value) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in capillary blood glucose between wholegrain products and reference in the 2-hour iPeak(0-120 min) (incremental maximum value) after the breakfast meal.
Postprandial Insulin iAUC(0-120 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in venous blood insulin between wholegrain products and reference in the total incremental area under the curve iAUC(0-120 min) after the standardized breakfast meal.
Postprandial Insulin Cmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in venous blood insulin between wholegrain products and reference in Cmax after the standardized breakfast meal.
Postprandial Insulin Tmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in venous blood insulin between wholegrain products and reference in Tmax after the standardized breakfast meal.
Fasting Insulin | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in fasting venous blood insulin the morning after consuming either wholegrain products or reference.
Postprandial insulin iAUC (0-60 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in venous blood insulin between wholegrain products and reference in the 1-hour incremental area under the curve iAUC(0-60 min) after the standardized breakfast meal.
Postprandial venous blood insulin 2-hour iPeak(0-120 min) (incremental maximum value) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in venous blood insulin between wholegrain products and reference in the 2-hour iPeak(0-120 min) (incremental maximum value) after the breakfast meal.

OTHER OUTCOMES:
Fasting GLP-1 | Outcome measures will be assessed just before the standardized meal is consumed.
  The change in fasting GLP-1 the morning after consuming either wholegrain products or reference.
GLP-1 iAUC(0-120 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in GLP-1 between wholegrain products and reference in the total incremental area under the curve iAUC(0-120 min) after the standardized breakfast meal.
GLP-1 iAUC(0-60 min) | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in GLP-1 between wholegrain products and reference in the1-hour incremental area under the curve iAUC(0-60 min) after the standardized breakfast meal.
GLP-1 Cmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The changein GLP-1 between wholegrain products and reference in Cmax after the standardized breakfast meal.
GLP-1 Tmax | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in GLP-1 between wholegrain products and reference in Tmax after the standardized breakfast meal.
Fasting PYY | Outcome measures will be assessed just before the standardized meal is consumed.
  The change in fasting PYY the morning after consuming either wholegrain products or reference.
PYY 2-hour mean concentration | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in PYY between the wholegrain products and the reference in the 2-hour mean concentration after the breakfast meal.
PYY 1-hour mean concentration | Outcome measures will be assessed just before and immediately after the standardized meal is consumed.
  The change in PYY between the wholegrain products and the reference in the 1-hour mean concentration after the breakfast meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Aventure AB, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No